CLINICAL TRIAL: NCT04641546
Title: Effectiveness of an Occupation-Based Intervention Compared With Therapeutic Exercise for Older Adults With Shoulder Osteoarthritis: A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Occupation-Based Intervention Compared With Therapeutic Exercise for Older Adults With Shoulder OA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bay Path University (Other)
Responsible Party: Principal Investigator, Kelli Cabrera, Principal Investigator, Bay Path University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BayPathU
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis Shoulder
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupation-Based Intervention + Therapeutic Exercise Intervention Group (Experimental): Sixty-minute occupational therapy sessions were completed two times a week for six weeks consisting of 30 minutes therapeutic exercise followed by 30 minutes of occupation-based intervention.
  Interventions: Procedure: Therapeutic Exercise; Procedure: Occupation-Based Intervention
- Therapeutic Exercise Control Group (Experimental): Sixty-minute occupational therapy sessions were completed two times a week for six weeks consisting of therapeutic exercise only.
  Interventions: Procedure: Therapeutic Exercise

INTERVENTIONS:
Procedure: Therapeutic Exercise — Passive range of motion (PROM), active-assistive range of motion (AAROM), active range of motion (AROM), and strengthening activities.
Procedure: Occupation-Based Intervention — Collecting and placing items in cabinets, washing windows and tables, and hanging clothes on a clothesline.
  Arms: Occupation-Based Intervention + Therapeutic Exercise Intervention Group

SUMMARY:
As a registered and licensed occupational therapist, I completed a six-week evidence based research study to determine the effects of occupation-based intervention and therapeutic exercises versus therapeutic exercises alone.

DETAILED DESCRIPTION:
Importance: There is a need for evidence to support occupation-based intervention (OBI) for older adults with shoulder osteoarthritis (OA).

Objective: To evaluate the effectiveness of OBI on function in older adults with shoulder OA compared to therapeutic exercise (TE).

Design: Randomized controlled trial. Six-week intervention. 1-week and 4-week follow-up.

Setting: Outpatient clinic. Participants: Ten older adults with diagnosis of shoulder OA via convenience sampling.

Intervention: Participants were seen two times/week for six weeks. The OBI group completed 30 minutes of TE followed by 30 minutes of OBI. The TE group completed 60 minutes of TE.

Outcome and Measures: Functional outcomes were assessed at pre-, 1-week post, and 4-weeks posttreatment using the QuickDASH as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of shoulder osteoarthritis (confirmed by physician examination or radiographic imaging)
* Aged 65 years or older

Exclusion Criteria:

* Previous shoulder injuries
* Acute pathology
* Previous shoulder surgery
* Current use of pain medication
* Inflammatory arthritis
* Upper extremity neuropathy or myopathy
* Current participation in a home exercise program
* Score of <18 on the Mini-Mental State Examination (MMSE)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) Baseline scores | Pre-Intervention
  To assess the impact of the intervention on physical function and symptoms of shoulder osteoarthritis.
  * Minimum Value: 0 (no disability)
  * Maximum Value: 100 (most severe disability)
  * Higher scores = Worse outcome (greater upper extremity dysfunction)
Change between Pre-Intervention and 1-week Post-Intervention Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) scores | 1-week Post-Intervention
  To assess the impact of the intervention on physical function and symptoms of shoulder osteoarthritis.
  * Minimum Value: 0 (no disability)
  * Maximum Value: 100 (most severe disability)
  * Higher scores = Worse outcome (greater upper extremity dysfunction)
Change between Pre-Intervention and 4-weeks Post-Intervention Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) scores | 4-weeks Post-Intervention
  To assess the impact of the intervention on physical function and symptoms of shoulder osteoarthritis.
  * Minimum Value: 0 (no disability)
  * Maximum Value: 100 (most severe disability)
  * Higher scores = Worse outcome (greater upper extremity dysfunction)
Change between 1-week and 4-weeks Post-Intervention Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) scores | 4-weeks Post-Intervention
  To assess the impact of the intervention on physical function and symptoms of shoulder osteoarthritis.
  * Minimum Value: 0 (no disability)
  * Maximum Value: 100 (most severe disability)
  * Higher scores = Worse outcome (greater upper extremity dysfunction)

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) Baseline Scores | Pre-Intervention
  To determine the effect of the intervention on participants' self-perception of occupational performance and satisfaction over time.
  * Minimum Value: 0
  * Maximum Value: 10
  * Higher scores = Better outcome (greater client-perceived changes in satisfaction and performance of daily occupations)
Change between Pre-Intervention and 1-week Post-Intervention Canadian Occupational Performance Measure (COPM) scores | 1-week Post-Intervention
  To determine the effect of the intervention on participants' self-perception of occupational performance and satisfaction over time.
  * Minimum Value: 0
  * Maximum Value: 10
  * Higher scores = Better outcome (greater client-perceived changes in satisfaction and performance of daily occupations)
Change between Pre-Intervention and 4-weeks Post-Intervention Canadian Occupational Performance Measure (COPM) scores | 4-weeks Post-Intervention
  To determine the effect of the intervention on participants' self-perception of occupational performance and satisfaction over time.
  * Minimum Value: 0
  * Maximum Value: 10
  * Higher scores = Better outcome (greater client-perceived changes in satisfaction and performance of daily occupations)
Change between 1-week and 4-weeks Post-Intervention Canadian Occupational Performance Measure (COPM) scores | 4-weeks Post-Intervention
  To determine the effect of the intervention on participants' self-perception of occupational performance and satisfaction over time.
  * Minimum Value: 0
  * Maximum Value: 10
  * Higher scores = Better outcome (greater client-perceived changes in satisfaction and performance of daily occupations)
Shoulder Range of Motion (ROM) Baseline Scores | Pre-Intervention
  Observing and grading ROM on a 3-point Likert scale to determine shoulder mobility and pain with movement.
  * Minimum Value: 0 (unable/no pain)
  * Maximum Value: 3 (full able/lots of pain)
  * Higher scores = Better outcome (fully ROM/no pain with ROM)
Change between Pre-Intervention and 1-week Shoulder Range of Motion (ROM) scores | 1-week Post-Intervention
  Observing and grading ROM on a 3-point Likert scale to determine shoulder mobility and pain with movement.
  * Minimum Value: 0 (unable/no pain)
  * Maximum Value: 3 (fully able/lots of pain)
  * Higher scores = Better outcome (full ROM/no pain with ROM)
Change between Pre-Intervention and 4-weeks Post-Intervention Shoulder Range of Motion (ROM) scores | 4-weeks Post-Intervention
  Observing and grading ROM on a 3-point Likert scale to determine shoulder mobility and pain with movement.
  * Minimum Value: 0 (unable/no pain)
  * Maximum Value: 3 (fully able/lots of pain)
  * Higher scores = Better outcome (full ROM/no pain with ROM)
Change between 1-week and 4-weeks Post-Intervention Shoulder Range of Motion (ROM) scores | 4-weeks Post-Intervention
  Observing and grading ROM on a 3-point Likert scale to determine shoulder mobility and pain with movement.
  * Minimum Value: 0 (unable/no pain)
  * Maximum Value: 3 (fully able/lots of pain)
  * Higher scores = Better outcome (full ROM/no pain with ROM)
Jamar Hand Dynamometer Baseline Scores | Pre-Intervention
  To measure grip strength.
  * Minimum Value: 0 pounds
  * Maximum Value: 200 pounds
  * Higher scores = Better outcome (increased grip strength)
Change between Pre-Intervention and 1-week Jamar Hand Dynamometer scores | 1-week Post-Intervention
  To measure grip strength.
  * Minimum Value: 0 pounds
  * Maximum Value: 200 pounds
  * Higher scores = Better outcome (increased grip strength)
Change between Pre-Intervention and 4-weeks Post-Intervention Jamar Hand Dynamometer scores | 4-weeks Post-Intervention
  To measure grip strength.
  * Minimum Value: 0 pounds
  * Maximum Value: 200 pounds
  * Higher scores = Better outcome (increased grip strength)
Change between 1-week and 4-weeks Post-Intervention Jamar Hand Dynamometer Scores | 4-weeks Post-Intervention
  To measure grip strength.
  * Minimum Value: 0 pounds
  * Maximum Value: 200 pounds
  * Higher scores = Better outcome (increased grip strength)
Numeric Pain Rating Scale (NPRS) Baseline Scores | Pre-Intervention
  To measure pain.
  * Minimum Value: 0 (no pain)
  * Maximum Value: 10 (worst possible pain)
  * Higher scores = Worse outcome (increased pain)
Change between Pre-Intervention and 1-week Numeric Pain Rating Scale (NPRS) Scores | 1-week Post-Intervention
  To measure pain.
  * Minimum Value: 0 (no pain)
  * Maximum Value: 10 (worst possible pain)
  * Higher scores = Worse outcome (increased pain)
Change between Pre-Intervention and 4-weeks Post-Intervention Numeric Pain Rating Scale (NPRS) Scores | 4-weeks Post-Intervention
  To measure pain.
  * Minimum Value: 0 (no pain)
  * Maximum Value: 10 (worst possible pain)
  * Higher scores = Worse outcome (increased pain)
Change between 1-week and 4-weeks Post-Intervention Numeric Pain Rating Scale (NPRS) scores | 4-weeks Post-Intervention
  To measure pain.
  * Minimum Value: 0 (no pain)
  * Maximum Value: 10 (worst possible pain)
  * Higher scores = Worse outcome (increased pain)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli A Cabrera, Principal Investigator — Bay Path University
Locations (1):
- Bay Path University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish research findings to the American Journal of Occupational Therapy (AJOT).
Supporting Information: Study Protocol, CSR
Time Frame: Within the next year

REFERENCES:
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Bull D, Tai Kie A, Hanusch B, Kulkarni R, Rees J, Rangan A. Is there sufficient evidence to support intervention to manage shoulder arthritis? Shoulder Elbow. 2016 Apr;8(2):77-89. doi: 10.1177/1758573215622385. Epub 2016 Jan 8. PMID 27583004
- [Background] Burner T, Abbott D, Huber K, Stout M, Fleming R, Wessel B, Massey E, Rosenthal A, Burns E. Shoulder symptoms and function in geriatric patients. J Geriatr Phys Ther. 2014 Oct-Dec;37(4):154-8. doi: 10.1519/JPT.0b013e3182abe7d6. PMID 24534849
- [Background] Che Daud AZ, Yau MK, Barnett F, Judd J, Jones RE, Muhammad Nawawi RF. Integration of occupation based intervention in hand injury rehabilitation: A Randomized Controlled Trial. J Hand Ther. 2016 Jan-Mar;29(1):30-40. doi: 10.1016/j.jht.2015.09.004. Epub 2015 Nov 6. PMID 26847318
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Marinko LN, Chacko JM, Dalton D, Chacko CC. The effectiveness of therapeutic exercise for painful shoulder conditions: a meta-analysis. J Shoulder Elbow Surg. 2011 Dec;20(8):1351-9. doi: 10.1016/j.jse.2011.05.013. Epub 2011 Sep 1. PMID 21889366
- [Background] McDonough CM, Jette AM. The contribution of osteoarthritis to functional limitations and disability. Clin Geriatr Med. 2010 Aug;26(3):387-99. doi: 10.1016/j.cger.2010.04.001. PMID 20699161
- [Background] Millett PJ, Gobezie R, Boykin RE. Shoulder osteoarthritis: diagnosis and management. Am Fam Physician. 2008 Sep 1;78(5):605-11. PMID 18788237
- [Background] Mushtaq S, Choudhary R, Scanzello CR. Non-surgical treatment of osteoarthritis-related pain in the elderly. Curr Rev Musculoskelet Med. 2011 Sep;4(3):113-22. doi: 10.1007/s12178-011-9084-9. PMID 21701816
- [Background] Weinstock-Zlotnick G, Mehta SP. A systematic review of the benefits of occupation-based intervention for patients with upper extremity musculoskeletal disorders. J Hand Ther. 2019 Apr-Jun;32(2):141-152. doi: 10.1016/j.jht.2018.04.001. Epub 2018 Jul 14. PMID 30017413

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT04641546/Prot_SAP_ICF_000.pdf